CLINICAL TRIAL: NCT00570154
Title: Pilot Study of Monocyte Biology in Insulin Sensitive, Resistant and Diabetic Subjects
Brief Title: Relation of White Blood Cell Function to Diabetes
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080028; 08-H-0028
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-10-19

CONDITIONS: Diabetes
Keywords: Mitochondrial Function in Monocytes; Macrophages and Diabetes or Insulin Resistance; Peripheral Blood Mononuclear Cells; Diabetes; Monocyte; Macrophages; Proteome; Type 2 Diabetes; Insulin Resistance; Insulin Sensitivity; Pre-Diabetes; Healthy Volunteer; HV
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

Patients who are pre-diabetic or have adult onset (type 2) diabetes have a significantly greater risk of developing heart, blood vessel, or kidney diseases.

Recent studies have shown that abnormalities in white blood cell function may increase the chances of developing insulin resistance, the underlying problem in diabetic or pre-diabetic patients.

Objectives:

To determine levels of insulin sensitivity in selected volunteers.

To compare the white blood cells of non-diabetic, pre-diabetic, and type 2 (adult onset) diabetic volunteers to evaluate possible differences in white blood cell function.

Eligibility:

Individuals between 21 and 60 years of age who (1) are non-diabetic, (2) are pre-diabetic (glucose intolerant or insulin resistant), or (3) have type 2 diabetes that is controlled by diet and/or medications other than insulin.

Design:

Evaluations before treatment:

* Blood tests, including screening procedures for blood-transmitted diseases such as hepatitis B and C, insulin sensitivity and glucose tolerance tests, and liver and kidney function tests.
* Pregnancy tests for women of childbearing age.

Two tests will be performed during the study period:

* Glucose tolerance test to determine how well the body uses glucose.
* Blood drawn to study white blood cells.

Participants will be financially compensated for the time spent during the study.

DETAILED DESCRIPTION:
Type II diabetes mellitus is rapidly becoming a global pandemic with a deleterious impact on cardiovascular morbidity and mortality. Understanding its pathophysiology is important for the development of future therapeutic interventions. Interestingly, mitochondrial dysfunction in skeletal muscle and adipose tissue are early events in the development of type II diabetes mellitus and are proposed to play a role in exacerbating insulin resistance. The genetic disruption of macrophage mitochondrial biology in preclinical studies results in the development of insulin resistance and concurrent mitochondrial dysfunction in peripheral tissue including skeletal muscle and the liver. Whether this disruption of mitochondrial function is evident in human mononuclear cells is unknown. We propose that the disruption of mitochondrial function in circulating cells may contribute to not only peripheral insulin resistance but may also evoke the myriad of vascular complications associated with diabetes.

To test these assumptions, we propose an initial proof of concept study to evaluate mitochondrial biology in circulating monocytes in normal volunteers, pre-diabetic and diabetic subjects to assess whether mitochondrial disruption/dysfunction evolves with the progression to type II diabetes. In parallel, gene expression and proteomic analysis will be performed to evaluate whether the development of insulin resistance and diabetes confers a specific modulation in the biological signature of monocytes with disease progression. To delineate these concepts we will evaluate study subjects' glucose tolerance and insulin sensitivity and draw blood to examine peripheral monocytes. Biological readouts will include: 1) the quantification of the mitochondrial genomic and electron transfer chain content; 2) the determination of mitochondrial reactive oxygen species capacity and defenses; 3) the pattern of monocyte differentiation and 4) the unbiased assessment of monocyte gene expression and proteome.

If the mitochondrial hypothesis is operational, this study will show that the mitochondrial disruption/dysfunction is a more generalized finding in type II diabetes. This would establish targeting the modification of mitochondrial function in various tissue/cell types as a novel strategy in the prevention and/or reversal of insulin resistance and diabetes.

ELIGIBILITY:
* INCLUSION CRITERIA (young groups)

Adults older than 21 years and less than 40 years

Subjects must either have:

Insulin sensitivity with a fasting blood glucose less than 100 mg/dl and a 2-hour post oral glucose tolerance test blood glucose less than 140 mg/dl

or

Insulin resistance as defined by a fasting blood sugar of greater than or equal to 100mg/dl but less than 125 mg/dl and/or a 2-hour post oral glucose tolerance test blood glucose greater than 140 mg/dl and less than 200 mg/dl.

Subject understands protocol and provides written, informed consent.

INCLUSION CRITERIA (middle age groups)

Adults greater than or equal to 40 years and less than or equal to 60 years

Subjects must either have:

Insulin sensitivity with a fasting blood glucose less than 100 mg/dl and a 2-hour post oral glucose tolerance test blood glucose less than 140 mg/dl

or

Insulin resistance as defined by a fasting blood sugar of greater than or equal to 100mg/dl but less than 125 mg/dl and/or a 2-hour post oral glucose tolerance test blood glucose greater than 140 mg/dl and less than 200 mg/dl.

or

Type II diabetes as defined by a fasting blood sugar of greater than 125 mg/dl and/or a 2-hour post oral glucose tolerance test blood glucose greater than 200 mg/dl if untreated and/or if subjects are on oral hypoglycemic agent therapy where the HbA1c is greater than 6.7 percent.

Subject understands protocol and provides written, informed consent.

EXCLUSION CRITERIA (all study volunteers and subjects)

Uncontrolled hypertension or therapy with a Beta-blocker

History of heart failure (or ejection fraction less than 55 percent by echocardiogram), unstable coronary artery disease or symptomatic peripheral arterial disease requiring changes in medication or medical intervention in the preceding 3 months.

Insulin-dependant diabetes mellitus or current use of thiazolidinediones

Women of childbearing age unless recent pregnancy test is negative and you are not breast feeding.

Serum creatinine greater than 2.5 mg/dl

Liver transaminase levels greater than 2.5 times upper limit of normal

History of cancer in the last 5 years

Active inflammatory disease, or infection, or abnormal white blood cell differential

Enrollment in any drug studies within the last 30 days

BMI greater than 35 for the middle age group and greater than 30 for the younger subjects

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2007-11-27; Primary Completion 2009-10-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barr EL, Zimmet PZ, Welborn TA, Jolley D, Magliano DJ, Dunstan DW, Cameron AJ, Dwyer T, Taylor HR, Tonkin AM, Wong TY, McNeil J, Shaw JE. Risk of cardiovascular and all-cause mortality in individuals with diabetes mellitus, impaired fasting glucose, and impaired glucose tolerance: the Australian Diabetes, Obesity, and Lifestyle Study (AusDiab). Circulation. 2007 Jul 10;116(2):151-7. doi: 10.1161/CIRCULATIONAHA.106.685628. Epub 2007 Jun 18. PMID 17576864
- [Background] Morino K, Petersen KF, Shulman GI. Molecular mechanisms of insulin resistance in humans and their potential links with mitochondrial dysfunction. Diabetes. 2006 Dec;55 Suppl 2(Suppl 2):S9-S15. doi: 10.2337/db06-S002. PMID 17130651
- [Background] Lowell BB, Shulman GI. Mitochondrial dysfunction and type 2 diabetes. Science. 2005 Jan 21;307(5708):384-7. doi: 10.1126/science.1104343. PMID 15662004